CLINICAL TRIAL: NCT04867642
Title: A First-In-Human, Randomized, Participant-Blind, Investigator-Blind, Placebo-Controlled, Single- and Multiple-Dose, Dose-Escalating Study Evaluating the Safety, Tolerability, and Pharmacokinetics of UCB0022 in Healthy Participants and Participants With Parkinson's Disease
Brief Title: A Study to Test the Safety, Tolerability, and Blood Levels of UCB0022 in Healthy Participants and Participants With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0091; 2020-003111-10 (EudraCT Number)
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Study Participants; Parkinson's Disease
Keywords: Healthy Study Participants; Parkinson's Disease; Phase 1; escalating cohorts; UCB0022
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The study consists of a crossover design part (Part A), two parts (Part B and Part C) with a parallel design and the open-label Part D.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a participant- and investigator-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A Sequence 1 (Experimental): Study participants randomized to Part A will receive single ascending doses of UCB0022 or placebo (PBO) at pre-specified time points during the Treatment Period of alternating cohorts in a crossover design.
  Interventions: Drug: UCB0022; Other: Placebo
- Part A Sequence 2 (Experimental): Study participants randomized to Part A will receive single ascending doses of UCB0022 or placebo (PBO) at pre-specified time points during the Treatment Period of alternating cohorts in a crossover design.
  Interventions: Drug: UCB0022; Other: Placebo
- Part B UCB0022 (Experimental): Study participants randomized to Part B will receive multiple ascending doses of UCB0022 at pre-specified time points during the Treatment Period of cohorts in a parallel design.
  Interventions: Drug: UCB0022
- Part B Placebo (Placebo Comparator): Study participants randomized to Part B will receive placebo (PBO) comparator at pre-specified time points during the Treatment Period of cohorts in a parallel design.
  Interventions: Other: Placebo
- Part C UCB0022 (Experimental): Study participants randomized to this cohort in Part C will receive fixed multiple doses of UCB0022 at pre-specified time points during the Treatment Period.
  Interventions: Drug: UCB0022
- Part C Placebo (Placebo Comparator): Study participants randomized to this cohort in Part C will receive placebo (PBO) comparator at pre-specified time points during the Treatment Period.
  Interventions: Other: Placebo
- Part D UCB0022 (Experimental): Study participants randomized to this cohort in Part D will receive a single dose of UCB0022 at a pre-specified time point during the Treatment Period.
  Interventions: Drug: UCB0022

INTERVENTIONS:
Drug: UCB0022 — Study participants will receive doses of UCB0022 in a pre-specified sequence during the Treatment Period of Part A, B, C and D.
  Arms: Part A Sequence 1; Part A Sequence 2; Part B UCB0022; Part C UCB0022; Part D UCB0022
Other: Placebo — Study participants will receive placebo comparator in a pre-specified sequence during the Treatment Period of Part A, B and C.
  Other Names: PBO
  Arms: Part A Sequence 1; Part A Sequence 2; Part B Placebo; Part C Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetic (PK) of UCB0022 and food effect.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive or 35 to 75 years for part C, at the time of signing the informed consent
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Study participant has a blood pressure (BP) and heart rate (HR) before the first dose, as determined by triplicate BP/HR measurements in a supine position, of mean systolic BP ranging between 90 and 130 millimeters of mercury (mmHg), mean diastolic BP ranging between 50 and 80 mmHg, and mean HR between 45 and 90 beats per minute (bpm)
* Participant has a body weight of at least 45 kg and body mass index (BMI) within the range 18 to 30 kg/m^2 (inclusive)
* Participants are male or female:
* A male participant must agree to use contraception as detailed in the protocol during the treatment period and for at least 7 days after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

Not a woman of childbearing potential (WOCBP) as defined in the protocol OR A WOCBP who agrees to follow the contraceptive guidance in the protocol during the Treatment Period and for at least 90 days after the last dose of study treatment

Part C only:

* Patient must have a documented history of idiopathic Parkinson's disease confirmed by a neurologist, and with no other atypical or secondary parkinsonism (eg, multiple-system atrophy, progressive supranuclear palsy, or evidence of drug-induced parkinsonism)
* Participants with Hoehn and Yahr Stages of 1 to 3 inclusive, (Hoehn and Yahr, 1967) at Screening when in the ON state
* Participants on stable dosage of all anti-Parkinsonian therapy for at least 30 days prior to first investigational medicinal product (IMP) administration (with the exception that MAO-B inhibitors that must be maintained at a stable level for at least 8 weeks prior), and it is anticipated that no changes will be needed during the course of the study
* Participant has a BP and HR at Screening, as determined by triplicate BP/HR measurements in a supine position, of mean systolic BP ranging between 90 and 140 mmHg, mean diastolic BP ranging between 50 and 90 mmHg, and a mean HR between 50 and 90 bpm

Exclusion Criteria:

* Participant has history or presence of cerebro/cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, psychiatric or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Participant has a high risk for cardiovascular accident based on family history or on laboratory test
* Participants with hypertension requiring medical treatment within 6 months before the Screening, or with clinically significant orthostatic hypotension
* Participant has a known hypersensitivity to any components of the study medication or comparative drugs (and/or an investigational device) as stated in this protocol
* Participant has a history of unexplained syncope or a family history of sudden death due to long QT syndrome
* Participant has active neoplastic disease or history within the past 5 years of screening visit except for basal cell or squamous epithelial carcinomas of the skin that have been treated with SOC. Study participant has a history of a major organ transplant or hematopoietic stem cell/marrow transplant
* Participant has past or intended use of over-the-counter or prescription medication including herbal medications within 2 weeks or 5 half-lives prior to dosing
* Participant has used hepatic enzyme-inducing drugs within 2 months prior to dosing
* Participant has alanine transaminase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.0x upper limit of normal (ULN)
* Participant has current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Participant has a current history of alcohol or drug use disorder within the last Y Statistical Manual of Mental Disorders Version 5 (DSM-5), within the last year
* Participant has any clinically relevant electrocardiogram (ECG) finding at the Screening Visit or at Baseline
* Participant has the presence of hepatitis B surface antigen (HBsAg) at Screening or within 3 months prior to dosing
* Participant has a positive hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention
* Participant has a positive human immunodeficiency virus (HIV) antibody test
* Participant has clinical signs and symptoms consistent with COVID-19 or had a positive Sars-Cov-2 test result within the last 4 weeks prior to dosing
* Active treatment or a history of glaucoma

Part C only:

* Participant with implantable intracranial stimulator or history of intracranial surgery
* Participant with documented diagnosis of dementia or a Montreal Cognitive Assessment (MoCA) score <26 at screening
* Participant with history of psychotic symptoms (including significant hallucinations) requiring treatment with an antipsychotic medication within the 12 months prior to Admission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent adverse events (TEAEs) | From Baseline (Day 1) to end of study Visit (up to Day 29 Part A) (up to Day 21 Part B and C)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A treatment-emergent adverse event is defined as any event not present prior to the initiation of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment.

SECONDARY OUTCOMES:
Maximum plasma concentration (cmax) for each single dose of UCB0022 in Part A | From Day 1 (predose) at predefined time points (up to Day 3)
  Cmax: Maximum plasma concentration for each pre-specified single dose in Part A
Time to maximum plasma concentration (tmax) for each single dose of UCB0022 in Part A | From Day 1 (predose) at predefined time points (up to Day 3)
  tmax: time to maximum plasma concentration for each single dose of UCB0022 in Part A
Area under the plasma concentration-time curve from time zero to infinity (AUC) for a each dose of UCB0022 in Part A | From Day 1 (predose) at predefined time points (up to Day 3)
  AUC (AUCinfinity): Area under the UCB0022 plasma concentration-time curve from time zero to infinity for a each dose in Part A
Maximum plasma concentration during a dosing interval through steady state (Cmax, ss) for each dose UCB0022 in Part B and C | From Day 1 (predose) at predefined time points (up to Day 16)
  Cmax, ss: Maximum plasma concentration during a dosing interval through steady state for each dose UCB0022 in Part B and Part C
Time to maximum plasma concentration during a dosing interval through steady state (tmax, ss) for each dose UCB0022 in Part B and C | From Day 1 (predose) at predefined time points (up to Day 16)
  tmax, ss: time to maximum plasma concentration during a dosing interval through steady state for each dose UCB0022 in Part B and Part C
Area under the plasma concentration-time curve at steady state (AUCtau) on Day 1 for a each dose of UCB0022 in Part B and C | From Day 1 (predose) at predefined time points to the last quantifiable concentration (Day 16)
  AUCtau: Area under the plasma concentration-time curve at steady state on Day 1 for a each dose of UCB0022 in Part B and C
Area under the plasma concentration-time curve at steady state (AUCtau) on Day 14 for a each dose of UCB0022 in Part B and C | From Day 1 (predose) at predefined time points to the last quantifiable concentration (Day 16)
  AUCtau: Area under the plasma concentration-time curve at steady state on Day 14 for a each dose of UCB0022 in Part B and C

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- UP0091 1, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.